Official Title: Developing Interoperable Tools for Anxiety and Depression Screening

NCT05864612

IRB Approval Date: 05/22/2024

Your epilepsy doctor has included questionnaires about your mood and anxiety as part of your clinic visit.

Taking part in this survey may involve providing information that you consider confidential or private. Depending upon how you answer these questions, the responses may be shared with your neurology provider. Some information you provide may be used for research. Careful efforts will be made to keep your information confidential. You will not lose any services, benefits, or rights if you choose not to participate in this voluntary survey.